CLINICAL TRIAL: NCT06798649
Title: Effect of Visual Presentation of Atherosclerotic Plaque on Modification of Arterial Hypertension One Year Postpartum in Women With a History of Adverse Pregnancy Outcomes, and Risk Customization With AI Prediction Algorithms: GESTA-COR Trial, a Prospective Randomised Clinical Trial
Brief Title: Effect of Visual Presentation of Atherosclerotic Plaque on Modification of Arterial Hypertension One Year Postpartum in Women With a History of Adverse Pregnancy Outcomes, and Risk Customization With AI Prediction Algorithms
Acronym: GESTA-COR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal-Infantil Vall d´Hebron Hospital (Other)
Responsible Party: Principal Investigator, Maria Goya, MD, PhD, Coordinator, Maternal-Infantil Vall d´Hebron Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hospital Vall d'Hebron; GESTA-COR TRIAL (Other: Vall d'Hebron Hospital)
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-01

CONDITIONS: Adverse Pregnancy Outcomes; Cardiovascular Diseases
Keywords: cardiovascular disease; vascular imaging; adverse pregnancy outocomes; preeclampsia; gestational diabetes; preterm birth; cardiovascular prevention; vascular health; clinical trial; health of women
MeSH Terms: conditions — Cardiovascular Diseases; Pre-Eclampsia; Diabetes, Gestational; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stantard management (No Intervention): Women with APOs RECEIVE standard health information but NO receive detailed vascular imaging results.
- Intervention group - images vision (Experimental): Women with APOs RECEIVE standard health information PLUS vascular imaging results.
  Interventions: Other: The intervention in the GESTACOR study involves providing detailed feedback from vascular imaging to women who have experienced adverse pregnancy outcomes (APOs).

INTERVENTIONS:
Other: The intervention in the GESTACOR study involves providing detailed feedback from vascular imaging to women who have experienced adverse pregnancy outcomes (APOs). — This is aimed at assessing whether such feedback can encourage the adoption of healthier lifestyles and enhance adherence to preventive treatments, thereby potentially reducing the incidence of postpartum hypertension and other cardiovascular diseases.
  Components of the Intervention:
  Vascular Imaging:
  Women in the intervention group undergo advanced vascular imaging using ultrasound technology to detect the presence of arterial plaques vs. no information about vascular images in the standard manag group.
  The images are analyzed to assess the extent of vascular health, focusing on areas typically affected by cardiovascular risks such as the carotid arteries.
  Feedback Delivery:
  Detailed results from the vascular imaging are provided to the participants in a comprehensible format by healthcare professionals specialized in cardiovascular health.
  This feedback session includes a thorough explanation of the findings, highlighting areas of concern and potential risks.
  Arms: Intervention group - images vision

SUMMARY:
The GESTA-COR study is a prospective, non-commercial, randomized clinical trial designed to evaluate the impact of detailed vascular imaging feedback on the management of cardiovascular health in women with a history of adverse pregnancy outcomes (APOs). The trial aims to determine if providing these women with detailed images of their vascular status can encourage the adoption of healthier lifestyles and adherence to preventive treatments, thereby potentially reducing the incidence of postpartum hypertension and other cardiovascular diseases.

This study involves two randomized groups:

Intervention Group (Randomized): Women with APOs receiving detailed vascular imaging results.

Standard Management Group (Randomized): Women with APOs who will continue receiving standard health information without vascular imaging results.

Participants will be monitored for 12 months postpartum, focusing on blood pressure levels, cardiovascular health indicators, and lifestyle changes.

DETAILED DESCRIPTION:
Detailed Description:

The GESTACOR study explores the proactive use of vascular imaging to improve cardiovascular health management in women who have experienced adverse pregnancy outcomes (APOs). This trial uniquely integrates advanced imaging techniques with traditional cardiovascular health assessments to evaluate the efficacy of visual feedback on health behaviour and management.

Methodology:

Participants are randomly assigned to two groups: one receiving detailed imaging feedback and the other receiving standard care without specific imaging results.

Vascular imaging involves state-of-the-art ultrasound techniques to detect arterial plaque, which could be indicative of heightened cardiovascular risk.

Over 12 months, participants undergo regular health assessments, including blood pressure monitoring, lipid profiling, and glucose testing, complemented by behavioural health evaluations to capture lifestyle modifications and adherence to prescribed medical regimens.

Expected Impacts:

The trial is structured to assess whether detailed feedback on vascular health can lead directly to better health outcomes through improved patient engagement and adherence to preventive measures.

Outcomes of this research may lead to new guidelines for postpartum women, particularly those with APOs, emphasizing early detection and intervention for cardiovascular risk factors.

Innovations and Advancements:

GESTA-COR is among the first studies to assess the direct impact of detailed vascular imaging feedback in a postpartum setting.

The study's design allows for the collection of significant data on the interplay between visual health information and patient-driven health management.

By focusing on a targeted female population traditionally underrepresented in cardiovascular research, GESTA-COR aims to fill a crucial gap in medical research and potential clinical practice, emphasizing gender-specific risk factors and tailored interventions. The findings could pave the way for integrated care approaches that significantly enhance long-term cardiovascular health in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older.
* History of one or more adverse pregnancy outcomes (APOs) such as preeclampsia, gestational diabetes, preterm birth before 37 weeks of gestation, or intrauterine growth restriction (fetal weight below the 10th percentile).

Exclusion Criteria:

* Women with a history of significant cardiovascular events such as myocardial infarction, angina, stroke, heart failure, recovered sudden death, or atrial fibrillation.
* Inability to provide informed consent.
* Women who do not meet the specific APO criteria set out for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant individuals after delivery
Enrollment: 318 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypertension rate after one year of the delivery | From the delivery until 1 year after delivery
  The primary objective of the GESTACOR study is to assess the effectiveness of detailed vascular imaging feedback in reducing the incidence of hypertension one year postpartum in women who have experienced adverse pregnancy outcomes (APOs). The study specifically targets the intervention group, providing them with detailed images of their vascular state to determine if this visual feedback can encourage adherence to healthier lifestyle choices and preventive healthcare measures. By directly linking these interventions with a reduction in postpartum hypertension, the study aims to establish a proactive approach to managing long-term cardiovascular risks in this population.

IPD SHARING:
Plan to Share IPD: Undecided